CLINICAL TRIAL: NCT03668665
Title: Influencing Wound Healing Through the Application of Hyaluronic Acid With Perfluorodecalin and Physalis Angulata Extract After Split Skin Removal From the Thigh - A Study in "Split Wound Design"
Acronym: Split Wound
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no approval by CA
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18-068
Record Dates: First submitted 2018-09-05; First posted 2018-09-12 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Wound Heal
Keywords: Split Skin Removal; Hyaloronic acid; Split Wound Design
MeSH Terms: interventions — perfluorodecalin

STUDY DESIGN:
Intervention Model Description: The wound is divided into two halves (top and bottom). During the in-patient stay, half of the split skin removal sites are treated with Ready Medical Post Treatment on the 1st, 4th and 7th postoperative days in addition to conventional treatment with moist dressings (Mepilex and Fixomull). The other half of the wound should only be treated with conventional dressings as a control. Half of those treated with Ready Medical Post Treatment receive a new dressing after each application.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The images taken from the wound as a progress control during the study should be evaluated anonymously by both the surgeon and the patient using the "Manchester Scar Scale" and the "Patient and Observer Scar Assessment Scale".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventionell Treatment (Active Comparator): After split skin removal, the wound is divided into 2 parts (=2 arms):
  1st half: conventional treatment with moist dressings (mepilex and fixomull)
  Interventions: Device: Conventionell Treatment
- Treatment with Ready Medical Post Treatment (Experimental): After split skin removal, the wound is divided into 2 parts (=2 arms):
  2nd half: conventional treatment with moist dressings (mepilex and fixomull) and additional treatment with ready medical post treatment
  Interventions: Drug: Ready Medical Post Treatment

INTERVENTIONS:
Drug: Ready Medical Post Treatment — Treatment of half of the wound with the product "ready medical post treatment" in addition to conventional treatment with moist dressings (Mepilex and Fixomull); on the 1st, 4th and 7th day after surgery, the product is applied to the wound and the dressing is changed
  Other Names: Hyaluronic acid combined with perfluorodecalin and Physalis angulata extract
  Arms: Treatment with Ready Medical Post Treatment
Device: Conventionell Treatment — Treatment of half of the wound with conventional moist dressings (Mepilex and Fixomull); a dressing change only takes place on the 7th day postoperatively
  Other Names: Wound treatment with moist dressings
  Arms: Conventionell Treatment

SUMMARY:
The study will use a split wound design to investigate whether secondary wound healing can be accelerated and improved by the application of hyaluronic acid combined with perfluorodecalin and Physalis angulata extract.

DETAILED DESCRIPTION:
In oral and maxillofacial surgery, split skin is regularly removed to cover secondary defects. These defects occur, for example, in tumor patients after the removal of microsurgical radialis or fibular grafts for defect coverage or reconstruction, since the skin cannot be primarily closed there.

Split skin is defined as a free skin graft made of epidermis and the upper parts of the dermis. The average thickness of the grafts is 0.2-0.8 mm. The thickness of the split skin determines the pigmentation structure and the quality of the graft. The thinner the split skin, the better the healing tendency and the less scar remains at the donor site. However, a disadvantage of thin split skin grafts is the stronger secondary shrinkage in the recipient region. Moderately thick grafts are hardly subject to scar shrinkage, but occasionally leave hypertrophic scars or keloids at the donor site. Split skin grafts with a thickness of 0.6-0.8 mm provide the best esthetic results, but have a poorer healing rate.

The split skin can be removed with a dermatome. The ventrolateral proximal thighs and the inside and outside of the upper arms are particularly suitable as donor regions.

In oral and maxillofacial surgery, a 0.4 mm thick split skin is usually removed from the ventrolateral thigh to cover the defect in the forearm or lower leg.

The requirement at the split skin removal site is rapid healing with complete re-epithelialization. To achieve this, wound management is currently left to the clinic itself, as there is no evidence-based standard care. The technical literature only recommends moist wound management and rare dressing changes.

A new product that promises faster healing and reduced scarring of these wounds is Ready Medical Post Treatment. This is an established preparation consisting of hyaluronic acid, perfluorodecalin and Physalis angulata extract. Studies have shown that both hyaluronic acid and perfluorodecalin can significantly improve the epithelialisation rate of wounds. The study will use a split wound design to investigate whether secondary wound healing can be accelerated and improved by the application of hyaluronic acid combined with perfluorodecalin and Physalis angulata extract.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-90 years
* Split skin removal at the thigh must be planned for the patients
* Adult patients who are mentally and physically able to understand the importance and scope of the study and to follow up the study staff
* Written informed consent before participating in the study

Exclusion Criteria:

* Patients suffering from a systemic disease (e.g. diabetes mellitus, anticoagulant therapy,...)
* Patients taking immunosuppressive drugs that may affect wound healing
* Patients suffering from skin diseases
* Pregnant and/or lactating women. Women of childbearing age should protect themselves from potential pregnancy by adequate contraception while participating in studies.
* Participation in a study may, at the investigator's discretion, present an unacceptable risk due to pre- or concomitant disease or the patient's general underlying condition.
* Underage, or older than 90 years
* Life span is less than six months
* There is a current or past medically relevant disease or treatment that could influence the evaluation of the study
* The patient has received a study medication within the last 30 days as part of another study
* Simultaneous participation in another clinical intervention study
* Expected lack of compliance
* Alcohol or drug abuse
* The patient is accommodated in an institution by official or court order
* Patients in a dependent relationship or employment relationship with the sponsor, investigator, or alternate investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Effect of Ready Medical Post Treatment on wound healing after split skin removal | 6.5 month
  Evaluation of the process control of wound healing (three-dimensional scans of the thigh) by surgeons and patients using questionnaire (wound assessment by "Patient and Observer Scar Assessment Scale")
  Patient and Observer Scar Assessment Scale: Vancouver Scar Scale, surface area; patient assessments of pain, itching, color, stiffness, thickness, relief (Score from 5 (best) to 50 (worse)
Effect of Ready Medical Post Treatment on wound healing after split skin removal | 6.5 month
  Evaluation of the process control of wound healing (three-dimensional scans of the thigh) by surgeons and patients using questionnaire (wound assessment by "Manchester Scar Scale")
  Manchester Scar Scale: VAS (Visual Analog Scale) plus scar color, skin texture, relationship to surrounding skin, texture, margins, size, multiplicity (Score from 5 (best) to 18 (worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral and maxillofacial surgery, University Hospital RWTH Aachen Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No